CLINICAL TRIAL: NCT00932529
Title: Use, Effects and Side-effects of Second-generation Antipsychotics in a Naturalistic Setting.
Acronym: BPP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Hugo A. Jørgensen, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSD-ID10591
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2003-12

CONDITIONS: Psychotic Disorders
Keywords: Antipsychotic drugs; Treatment effectiveness; Randomized controlled trial
MeSH Terms: conditions — Psychotic Disorders | interventions — Olanzapine; Quetiapine Fumarate; Risperidone; ziprasidone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Olanzapine (Active Comparator)
  Interventions: Drug: Olanzapine; Drug: Quetiapine; Drug: Ziprasidone
- Quetiapine (Active Comparator)
  Interventions: Drug: Olanzapine; Drug: Risperidone; Drug: Ziprasidone
- Risperidone (Active Comparator)
  Interventions: Drug: Olanzapine; Drug: Ziprasidone
- Ziprasidone (Active Comparator)
  Interventions: Drug: Olanzapine; Drug: Ziprasidone

INTERVENTIONS:
Drug: Olanzapine — Olanzapine tablets 2.5mg - 20 mg per day once daily, or at the treating clinicians discretion
  Other Names: Zyprexa
Drug: Quetiapine — Tablets, 25 mg-800 mg given twice daily, or at the treating clinicians discretion.
  Other Names: Seroquel
  Arms: Olanzapine
Drug: Risperidone — Tablets, 1mg-6mg per day, once or twice daily, or at the treating clinicians discretion.
  Other Names: Risperdal
  Arms: Quetiapine
Drug: Ziprasidone — Tablets, 20mg - 160 mg twice daily, or at the treating clinicians discretion
  Other Names: Zeldox, Geodon

SUMMARY:
Despite different pharmacological properties, the scientific evidence is inconclusive regarding which of the first-line second generation antipsychotics (SGAs) should be preferred for the individual patient suffering from psychosis. The limitations of the evidence base may be related to the highly selected samples, short duration, and rigid experimental designs of most randomized clinical trials of efficacy. Moreover a high proportion of the clinical trials are drug company sponsored which could introduce funding bias. The purpose of this non-commercially funded study is to investigate whether effectiveness differences exist among the first-line SGAs olanzapine, quetiapine, risperidone, and ziprasidone when the drugs are used in a representative clinical setting. Eligible patients are those admitted to hospital for acute psychosis and candidates for oral antipsychotic treatment. The investigators hypothesise that in the naturalistic setting of every-day clinical practice and in a diverse sample representative of most patients admitted for symptoms of acute psychosis, differential effectiveness among the SGAs could be disclosed when the patients are followed for up to 2 years. This could deliver valuable information regarding which SGA should be the starting antipsychotic drug in order to facilitate the most beneficial outcome.

ELIGIBILITY:
Inclusion Criteria:

* Psychosis
* Must be able to use oral antipsychotic drugs

Exclusion Criteria:

* Mania
* Unable to cooperate with the assessments
* Unable to understand Norwegian language
* Candidates for electroconvulsive therapy
* Use of Clozapine at admittance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2003-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Reduction of PANSS total score | Admission, discharge/ 6 weeks if not discharged, 3, 6, 12, 24 months after admittance.

SECONDARY OUTCOMES:
Tolerability | Discharge/ after 6 weeks if not discharged, 3, 6, 12, 24 months after discharge
Time until initial drug discontinuation | Up to 24 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Division of Psychiatry, Bergen, Sandviken, Norway

REFERENCES:
- [Derived] Bjarke J, Sinkeviciute I, Kroken RA, Loberg EM, Jorgensen HA, Johnsen E, Gjestad R. Different response patterns in hallucinations and delusions to antipsychotic treatment. Nord J Psychiatry. 2020 Oct;74(7):497-504. doi: 10.1080/08039488.2020.1745273. Epub 2020 Apr 3. PMID 32242498
- [Derived] Kjelby E, Gjestad R, Sinkeviciute I, Kroken RA, Loberg EM, Jorgensen HA, Johnsen E. Trajectories of depressive symptoms in the acute phase of psychosis: Implications for treatment. J Psychiatr Res. 2018 Aug;103:219-228. doi: 10.1016/j.jpsychires.2018.06.003. Epub 2018 Jun 2. PMID 29890508
- [Derived] Johnsen E, Fathian F, Kroken RA, Steen VM, Jorgensen HA, Gjestad R, Loberg EM. The serum level of C-reactive protein (CRP) is associated with cognitive performance in acute phase psychosis. BMC Psychiatry. 2016 Mar 14;16:60. doi: 10.1186/s12888-016-0769-x. PMID 26973142
- [Derived] Kjelby E, Sinkeviciute I, Gjestad R, Kroken RA, Loberg EM, Jorgensen HA, Hugdahl K, Johnsen E. Suicidality in schizophrenia spectrum disorders: the relationship to hallucinations and persecutory delusions. Eur Psychiatry. 2015 Oct;30(7):830-6. doi: 10.1016/j.eurpsy.2015.07.003. Epub 2015 Sep 25. PMID 26443050
- [Derived] Johnsen E, Aanesen K, Sriskandarajah S, Kroken RA, Loberg EM, Jorgensen HA. QTc Prolongation in Patients Acutely Admitted to Hospital for Psychosis and Treated with Second Generation Antipsychotics. Schizophr Res Treatment. 2013;2013:375020. doi: 10.1155/2013/375020. Epub 2013 Dec 31. PMID 24490070
- [Derived] Johnsen E, Sinkeviciute I, Loberg EM, Kroken RA, Hugdahl K, Jorgensen HA. Hallucinations in acutely admitted patients with psychosis, and effectiveness of risperidone, olanzapine, quetiapine, and ziprasidone: a pragmatic, randomized study. BMC Psychiatry. 2013 Sep 30;13:241. doi: 10.1186/1471-244X-13-241. PMID 24079855
- [Derived] Kjelby E, Jorgensen HA, Kroken RA, Loberg EM, Johnsen E. Anti-depressive effectiveness of olanzapine, quetiapine, risperidone and ziprasidone: a pragmatic, randomized trial. BMC Psychiatry. 2011 Aug 31;11:145. doi: 10.1186/1471-244X-11-145. PMID 21884578
- [Derived] Johnsen E, Gjestad R, Kroken RA, Mellesdal L, Loberg EM, Jorgensen HA. Cardiovascular risk in patients admitted for psychosis compared with findings from a population-based study. Nord J Psychiatry. 2011 Jun;65(3):192-202. doi: 10.3109/08039488.2010.522729. Epub 2010 Sep 29. PMID 20879830
- [Derived] Johnsen E, Kroken RA, Wentzel-Larsen T, Jorgensen HA. Effectiveness of second-generation antipsychotics: a naturalistic, randomized comparison of olanzapine, quetiapine, risperidone, and ziprasidone. BMC Psychiatry. 2010 Mar 24;10:26. doi: 10.1186/1471-244X-10-26. PMID 20334680